CLINICAL TRIAL: NCT03170219
Title: Subcutaneous Furosemide in Acute Decompensated Heart Failure: The SUBQ-HF Study
Acronym: SUBQ-HF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Adrian Hernandez (Other)
Responsible Party: Sponsor-Investigator, Adrian Hernandez, HFN Coordinating Center PI, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00070619
Record Dates: First submitted 2017-05-06; First posted 2017-05-30 (Actual); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Acute Heart Failure; Decompensated Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Subcutaneous Furosemide and sc2wear device (Experimental): Subjects will receive device training and study materials (SQ pump device and up to a 7 day supply of SQ furosemide vials) on the day of randomization (study day 0) and discharged within 24 hours. Subjects will be discharged with planned treatment of 80 mg subcutaneous furosemide injection over 5-hours either QD or BID, depending on anticipated diuretic requirements.
  Interventions: Combination Product: subcutaneous furosemide and sc2wear device
- Usual Care (No Intervention): Subjects randomized to usual care will continue to receive inpatient therapy, eventual transition to oral diuretics, and discharge and post discharge care as per the discretion of the treating clinician and standard treatment guidelines.

INTERVENTIONS:
Combination Product: subcutaneous furosemide and sc2wear device — subcutaneous furosemide administered via sc2wear device vs. standard of care
  Arms: Subcutaneous Furosemide and sc2wear device

SUMMARY:
To determine if a strategy of early discharge using a novel subcutaneous delivery system for parenteral furosemide can improve clinical outcomes within 30 days of randomization (days alive and outside the hospital) compared to usual care.

DETAILED DESCRIPTION:
SUBQ-HF is a multicenter clinical trial of selected AHF patients with persistent congestion. This study will evaluate a strategy of early discharge (pathway 1) or admission avoidance (pathway 2) with daily SQ furosemide compared to usual care in a population who have objective evidence of persistent congestion requiring ongoing parenteral diuretics. This will be an unblinded, randomized, controlled study of approximately 300 evaluable patients. Eligible patients will be randomized (1:1) to either:

Usual care strategy, during which patients will have continued inpatient treatment and discharge follow-up as per usual standard of care plus a Day 7 phone call and Day 30 study visit.

or

Subcutaneous strategy, in which patients will be discharged home within 24 hours of randomization (pathway 1) or sent home from clinic or ED to receive furosemide with the SQ pump for 1-7 days (based on clinical response) plus a Day 7 and Day 30 visit.

Subcutaneous furosemide/early discharge strategy:

Subjects will receive device training and study materials (SQ pump device and up to a 7 day supply of SQ furosemide vials) on the day of randomization (study day 0) and discharged within 24 hours. Training will include instruction on daily weights and dyspnea numerical rating for symptoms. Scales will be provided to subjects. Subjects will be discharged with planned treatment of 80 mg SQ furosemide injection over 5-hours either QD or BID, depending on anticipated diuretic requirements. If there are unanticipated delays in discharge after randomization, subjects will continue with their assigned therapy and assessments in the hospital. Discharged subjects will receive a phone contact from study team on D1, D3, and D5 in order to assess adequacy of diuresis, persistence of congestion, and planned duration, dose of ongoing SQ therapy (see Appendix for guidelines on adjusting therapy) and adverse events. Additional clinical contact (additional phone contacts or clinical visits) may be performed if felt clinically indicated by the study team or clinical provider. All subjects will have assessment of electrolytes and renal function by protocol 2 days post discharge. More frequent electrolyte monitoring can be performed at the discretion of the study team or clinical provider as clinically indicated. Patients receiving the SQ pump for outpatient use should be prescribed a supplementation regimen based on electrolyte supplementation needs in the hospital with IV diuretic therapy. The duration of subcutaneous therapy will be planned for 1-7 days depending on clinical response. Dose and frequency of oral diuretics once SQ therapy is completed will be per the discretion of the treating physician.

Usual care strategy:

Subjects randomized to usual care will continue to receive inpatient therapy, eventual transition to oral diuretics, and discharge and post discharge care as per the discretion of the treating clinician and standard treatment guidelines. In addition, they will have a Day 7 study phone call and a Day 30 study visit.

ELIGIBILITY:
Inclusion Criteria for Pathway 1 (patients hospitalized with acute heart failure)

1. Age >18 years
2. Willingness and ability to provide informed consent
3. Hospitalization for AHF with at least 1 symptom (dyspnea, orthopnea, or edema) AND 1 sign (rales on auscultation, peripheral edema, ascites, pulmonary vascular congestion on chest radiography, BNP > 250 ng/mL or NTproBNP > 1000 ng/mL) of congestion
4. Persistent congestion defined by the presence of at least 2 or more of the following at the time of consent:

   1. Peripheral edema
   2. Rales
   3. Elevated JVP
   4. Ascites
   5. BNP > 250 ng/mL or NTproBNP > 1000 ng/mL during index hospitalization
   6. Orthopnea
5. Total anticipated daily IV furosemide dose (at time of screening) >80-240 mg (or equivalent)/day
6. Anticipated need for at least 24 more hours of parenteral diuretic therapy

Exclusion Criteria for Pathway 1

1. Severe renal dysfunction (eGFR< 20 ml/min/1.73m2) within 24 hours of enrollment
2. Requirement for inotropes (other than digoxin) or mechanical support during hospitalization
3. Clinically significant electrical instability during hospitalization
4. Anticipated need for ongoing intravenous therapies beyond diuretics (electrolyte repletion, vasodilators, antibiotics, etc.)
5. Planned discharge to location other than home (e.g., hospice, skilled nursing facility, etc.)
6. Anticipated cardiac transplantation or left ventricular assist device within the next 30 days
7. Primary hypertrophic cardiomyopathy, infiltrative cardiomyopathy, acute myocarditis, constrictive pericarditis or tamponade
8. Known or anticipated pregnancy in the next 30 days
9. Prior use of a subcutaneous furosemide pump or current use of any subcutaneous pump, on-body infusion devices or patients who give regimented injections at the intended site of the furosemide infusion device.
10. Other psychosocial or physical barriers to following the protocol and using SQ pump device outside the hospital setting
11. Known allergy to furosemide
12. Known sensitivity or allergy to medical adhesive tape
13. Enrollment or planned enrollment in another therapeutic clinical trial in next 3 months
14. Presentation is for indication other than CHF

Inclusion Criteria for Pathway 2 (Outpatients with heart failure presenting with volume overload necessitating treatment with parenteral loop diuretics)

1. Age >18 years
2. Willingness and ability to provide informed consent
3. HF now presenting with volume overload defined by the presence of at least 2 or more of the following at the time of consent:

   1. Peripheral edema
   2. Rales
   3. Elevated JVP
   4. Ascites
   5. BNP > 250 ng/mL or NTproBNP > 1000 ng/mL during this episode of decompensation
   6. Orthopnea
4. Need for parenteral furosemide with an estimated SQ furosemide requirement between 80-240 mg/day
5. Anticipated need for at least 24 hours of parenteral diuretic therapy

Exclusion Criteria for Pathway 2

1. Severe renal dysfunction (eGFR< 20 ml/min/1.73m2) within 24 hours of enrollment
2. Anticipated need for inotropes (other than digoxin) or mechanical support to treat current episode of decompensation
3. Clinically significant electrical instability requiring hospitalization
4. Anticipated need for ongoing intravenous therapies beyond diuretics (electrolyte repletion, vasodilators, antibiotics, etc.)
5. Residence at location other than home (e.g., hospice, skilled nursing facility, etc.)
6. Anticipated cardiac transplantation or left ventricular assist device within the next 30 days
7. Primary hypertrophic cardiomyopathy, infiltrative cardiomyopathy, acute myocarditis, constrictive pericarditis or tamponade
8. Known or anticipated pregnancy in the next 30 days
9. Prior use of a subcutaneous furosemide pump or current use of any subcutaneous pump, on-body infusion devices or patients who give regimented injections at the intended site of the furosemide infusion device.
10. Other psychosocial or physical barriers to following the protocol and using SQ pump device outside the hospital setting
11. Known allergy to furosemide
12. Known sensitivity or allergy to medical adhesive tape
13. Enrollment or planned enrollment in another therapeutic clinical trial in next 3 months.
14. Presentation is for indication other than CHF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hernandez, MD, Principal Investigator — Duke University; Eugene Braunwald, MD, Study Chair — Harvard University
Locations (16):
- United States (16):
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Stony Brook University Medical Center, Stony Brook, New York
  - Duke University, Durham, North Carolina
  - University Hospitals- Case Medical Center, Cleveland, Ohio
  - Metro Health System, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvaina, Philadelphia, Pennsylvania
  - University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subcutaneous Furosemide and sc2wear Device | Usual Care
Started | 7 | 4
Completed | 7 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subcutaneous Furosemide and sc2wear Device | Usual Care | Total
Number analyzed (Participants) | 7 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (15.2) | 64.3 (6.4) | 62.2 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 4 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Patient Safety Measured by Serious Adverse Events
Description: measured by serious adverse events
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Furosemide and sc2wear Device | Usual Care
Number analyzed (Participants) | 7 | 4
Participants | 0 | 0

2. Secondary Outcome: Composite Safety Endpoint of Death, Sustained Ventricular Arrhythmias, and Severe Hypokalemia
Time Frame: 30 days
Population: Data not collected.
Arm/Group | Subcutaneous Furosemide and sc2wear Device | Usual Care
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Medical Costs From Randomization Through 30 Days
Time Frame: 30 days
Population: Data not collected.
Arm/Group | Subcutaneous Furosemide and sc2wear Device | Usual Care
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Days Alive and Outside the Hospital Through 14 Days
Time Frame: 14 days
Population: Data not collected.
Arm/Group | Subcutaneous Furosemide and sc2wear Device | Usual Care
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: 30 Day Heart Failure Readmission
Time Frame: 30 days
Population: Data not collected.
Arm/Group | Subcutaneous Furosemide and sc2wear Device | Usual Care
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: 30 Day ED Visit for Heart Failure
Time Frame: 30 days
Population: Data not collected.
Arm/Group | Subcutaneous Furosemide and sc2wear Device | Usual Care
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Death at 30 Days
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Furosemide and sc2wear Device | Usual Care
Number analyzed (Participants) | 7 | 4
Participants | 0 | 0

8. Secondary Outcome: Change in Breathlessness Through Day 7
Description: On a 0-10 scale of breathlessness
Time Frame: 7 days
Population: Data not collected.
Arm/Group | Subcutaneous Furosemide and sc2wear Device | Usual Care
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Renal Function Using eGFR Baseline to 30 Days
Time Frame: 30 days
Population: Data not collected.
Arm/Group | Subcutaneous Furosemide and sc2wear Device | Usual Care
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in NT Pro BNP From Baseline to 30 Days
Time Frame: 30 days
Population: Data not collected.
Arm/Group | Subcutaneous Furosemide and sc2wear Device | Usual Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Time of consent to day 30
Arm/Group | Subcutaneous Furosemide and sc2wear Device | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/4
Other Adverse Events (participants affected / at risk) | 3/7 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subcutaneous Furosemide and sc2wear Device (N=7) | Usual Care (N=4)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Transferrin Saturation Decreased (Investigations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT03170219/Prot_SAP_000.pdf